CLINICAL TRIAL: NCT01453205
Title: A Phase 2 Randomized Open-label Study of MEDI-551 in Adults With Relapsed or Refractory DLBCL
Brief Title: A Phase 2, Multicenter, Randomized, Open-label Study of MEDI-551 in Adults With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI-551-1088
Record Dates: First submitted 2011-10-03; First posted 2011-10-17 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma, Non-Hodgkin's Lymphoma, Diffuse Large B-Cell Lymphoma, DLBCL, B-Cell Malignancy, anti-CD19, monoclonal antibody, second line, ASCT, Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Non-Hodgkin | interventions — inebilizumab; Rituximab; Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rituximab+ ICE/DHAP (Active Comparator): Participants will receive Rituximab in combination with ifosfamide + carboplatin + etoposide (ICE) or dexamethasone + cisplatin + cytarabine (DHAP) for 3 cycles (21-day cycles) and will followed until end of the study (36 months after the date of randomization for last participant, or date the sponsor stops the trial, whichever occurs first). Rituximab (375 mg/m^2) will be administered intravenous (IV) on 2 days before the start of Cycle 1 and on Day 1 of each cycle. After completion of rituximab, IV infusion of ICE as: ifosfamide 5 g/ m^2 continuously for 24 hours with mesna on Day 2; carboplatin AUC=5 mg/mL x min (800 mg maximum) on Day 2; etoposide 100 mg/ m^2 on Days 1, 2, and 3 in 21-day cycles. After completion of rituximab, IV infusion of DHAP as: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m^2 continuously for 24 hours on Day 1; cytarabine 2 g/m^2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
  Interventions: Drug: Rituximab; Drug: ICE; Drug: DHAP; Procedure: Autologous Stem Cell Transplant (ASCT)
- MEDI-551 2 mg/kg + ICE/DHAP (Experimental): Participants will receive MEDI-551 (2 mg/kg) in combination with ICE or DHAP for 3 cycles (21-day cycles) and will be followed until end of the study (36 months after the date of randomization for last participant, or date the sponsor stops the trial, whichever occurs first). MEDI-551 (2 mg/kg) will be administered IV on 7 days before the start of Cycle 1 and on Day 1 of each cycle. After completion of MEDI-551, IV infusion of ICE as: ifosfamide 5 g/ m^2 continuously for 24 hours with mesna on Day 2; carboplatin AUC=5 mg/mL x min (800 mg maximum) on Day 2; etoposide 100 mg/ m^2 on Days 1, 2, and 3 in 21-day cycles. After completion of MEDI-551, IV infusion of DHAP as: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m^2 continuously for 24 hours on Day 1; cytarabine 2 g/m^2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
  Interventions: Drug: MEDI-551 2 mg/kg; Drug: ICE; Drug: DHAP; Procedure: Autologous Stem Cell Transplant (ASCT)
- MEDI-551 4 mg/kg + ICE/DHAP (Experimental): Participants will receive MEDI-551 (4 mg/kg) in combination with ICE or DHAP for 3 cycles (21-day cycles) and will be followed until end of the study (36 months after the date of randomization for last participant, or date the sponsor stops the trial, whichever occurs first). MEDI-551 (4 mg/kg) will be administered IV on 7 days before the start of Cycle 1 and on Day 1 of each cycle. After completion of MEDI-551, IV infusion of ICE as: ifosfamide 5 g/ m^2 continuously for 24 hours with mesna on Day 2; carboplatin AUC=5 mg/mL x min (800 mg maximum) on Day 2; etoposide 100 mg/ m^2 on Days 1, 2, and 3 in 21-day cycles. After completion of MEDI-551, IV infusion of DHAP as: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m^2 continuously for 24 hours on Day 1; cytarabine 2 g/m^2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
  Interventions: Drug: ICE; Drug: DHAP; Procedure: Autologous Stem Cell Transplant (ASCT); Drug: MEDI-551 4 mg/kg

INTERVENTIONS:
Drug: MEDI-551 2 mg/kg — MEDI-551 at the assigned dose will be administered via Intravenous (IV) infusion. Subjects will receive 3 cycles of M-ICE or M-DHAP unless CR is achieved at the end of Cycle 2, disease progression is noted at the end of Cycle 2, or a significant/serious drug related toxicity occurs (as per the opinion of the investigator).
  Other Names: Inebilizumab
  Arms: MEDI-551 2 mg/kg + ICE/DHAP
Drug: Rituximab — Rituximab at 375 mg/m2 will be administered via IV infusion 2 days before the start of Cycle 1 and on Day 1 of each cycle. The infusion time for rituximab will be 50 400 mg/hr, depending on subject's tolerance. Subjects will receive 3 cycles of Rituximab with Ice (R ICE) or Rituximab with DHAP (R-DHAP) unless CR is achieved at the end of Cycle 2, disease progression is noted at the end of Cycle 2, or a significant/serious drug related toxicity occurs (as per the opinion of the investigator).
  Other Names: Rituxan; MabThera
  Arms: Rituximab+ ICE/DHAP
Drug: ICE — ICE will be administered via IV infusion as follows: ifosfamide 5 g/m2 continuously for 24 hours with mesna on Days 2 and 3; carboplatin AUC=5 mg/mL x min [800 mg maximum) on Day 2; etoposide 100 mg/m2 on Days 1, 2, and 3) in 21-day cycles.
Drug: DHAP — DHAP will be administered via IV infusion as follows: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m2 continuously for 24 hours on Day 1 of dosing cycle; cytarabine 2 g/m2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
Procedure: Autologous Stem Cell Transplant (ASCT) — Subjects who achieve CR or PR will undergo stem cell harvest and autologous stem cell transplantation (ASCT) following standard institutional protocols.
Drug: MEDI-551 4 mg/kg — MEDI-551 at the assigned dose will be administered via Intravenous (IV) infusion. Subjects will receive 3 cycles of M-ICE or M-DHAP unless CR is achieved at the end of Cycle 2, disease progression is noted at the end of Cycle 2, or a significant/serious drug related toxicity occurs (as per the opinion of the investigator).
  Other Names: Inebilizumab
  Arms: MEDI-551 4 mg/kg + ICE/DHAP

SUMMARY:
The overall purpose of the study is to determine if MEDI-551, when used in combination with salvage chemotherapy, Ifosfamide-carboplatin-etoposide (ICE) or Dexamethasone-cytarabine (DHAP) in patients with relapsed or refractory DLBCL who are eligible for Autologous Stem Cell Transplant (ASCT), has superior efficacy compared to rituximab in the same population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aggressive B-cell DLBCL, including FL transforming to DLBCL & Grade III FL
* Relapsed from or refractory to at least one treatment containing rituximab or another anti-CD20 based immunotherapy combined with anthracycline- or anthracenedione-based chemotherapy
* Eligible for ASCT
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of ≥ 12 weeks
* Adequate hematological function

Exclusion Criteria:

* Any chemotherapy, radiotherapy, immunotherapy, biologic, investigational or hormonal therapy for treatment of lymphoma within 28 days prior to treatment
* Previous cancer therapy for DLBCL other than anthracycline- or anthracenedione based chemoimmunotherapy, monotherapy rituximab prior to first line therapy and/or as a maintenance therapy, or limited field radiotherapy
* Prior autologous or allogeneic SCT
* New York Heart Association ≥ Class II congestive heart failure; Clinically significant abnormality on ECG
* History of other invasive malignancy within 5 years except for localized/in situ, carcinomas such as cervical carcinoma in situ.
* Evidence of active infection
* Documented current central nervous system involvement by leukemia or lymphoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (74):
- United States (28):
  - Research Site, Birmingham, Alabama
  - Research Site, Burbank, California
  - Research Site, Palm Springs, California
  - Research Site, Sylmar, California
  - Research Site, Atlanta, Georgia
  - Research Site, Westwood, Kansas
  - Research Site, Hazard, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, Fargo, North Dakota
  - Research Site, Dayton, Ohio
  - Research Site, Newark, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Canada (3):
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Greenfield Park, Quebec
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- France (7):
  - Research Site, Bordeaux
  - Research Site, Le Mans
  - Research Site, Libourne
  - Research Site, Marseille
  - Research Site, Pessac
  - Research Site, Rouen
  - Research Site, Tours
- Germany (6):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Tübingen
  - Research Site, Würzburg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kaposvár
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- Poland (2):
  - Research Site, Gdynia
  - Research Site, Lublin
- Russia (2):
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
- Spain (12):
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, San Sebastián de los Reyes
  - Research Site, Seville
  - Research Site, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Izmir
  - Research Site, Kurupelit
  - Research Site, Malatya
  - Research Site, Talas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 27Feb2012 to 17Jun2016.
Pre-assignment Details: A total of 256 participants were screened, of which 187 participants were randomized in the study.
Groups:
- Rituximab+ ICE/DHAP: Participants received Rituximab in combination with ifosfamide + carboplatin + etoposide (ICE) or dexamethasone + cisplatin + cytarabine (DHAP) for 3 cycles (21-day cycles) and were followed until end of the study (36 months after the date of randomization for last participant, or date the sponsor stops the trial, whichever occurs first). Rituximab (375 mg/m^2) was administered intravenous (IV) on 2 days before the start of Cycle 1 and on Day 1 of each cycle. After completion of rituximab, IV infusion of ICE as: ifosfamide 5 g/ m^2 continuously for 24 hours with mesna on Day 2; carboplatin AUC=5 mg/mL x min (800 mg maximum) on Day 2; etoposide 100 mg/ m^2 on Days 1, 2, and 3 in 21-day cycles. After completion of rituximab, IV infusion of DHAP as: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m^2 continuously for 24 hours on Day 1; cytarabine 2 g/m^2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
- MEDI-551 2 mg/kg + ICE/DHAP: Participants received MEDI-551 (2 mg/kg) in combination with ICE or DHAP for 3 cycles (21-day cycles) and were followed until end of the study (36 months after the date of randomization for last participant, or date the sponsor stops the trial, whichever occurs first). MEDI-551 (2 mg/kg) was administered IV on 7 days before the start of Cycle 1 and on Day 1 of each cycle. After completion of MEDI-551, IV infusion of ICE as: ifosfamide 5 g/ m^2 continuously for 24 hours with mesna on Day 2; carboplatin AUC=5 mg/mL x min (800 mg maximum) on Day 2; etoposide 100 mg/ m^2 on Days 1, 2, and 3 in 21-day cycles. After completion of MEDI-551, IV infusion of DHAP as: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m^2 continuously for 24 hours on Day 1; cytarabine 2 g/m^2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
- MEDI-551 4 mg/kg + ICE/DHAP: Participants received MEDI-551 (4 mg/kg) in combination with ICE or DHAP for 3 cycles (21-day cycles) and were followed until end of the study (36 months after the date of randomization for last participant, or date the sponsor stops the trial, whichever occurs first). MEDI-551 (4 mg/kg) was administered IV on 7 days before the start of Cycle 1 and on Day 1 of each cycle. After completion of MEDI-551, IV infusion of ICE as: ifosfamide 5 g/ m^2 continuously for 24 hours with mesna on Day 2; carboplatin AUC=5 mg/mL x min (800 mg maximum) on Day 2; etoposide 100 mg/ m^2 on Days 1, 2, and 3 in 21-day cycles. After completion of MEDI-551, IV infusion of DHAP as: dexamethasone 40 mg on Days 1, 2, 3, and 4; cisplatin 100 mg/m^2 continuously for 24 hours on Day 1; cytarabine 2 g/m^2 in 3-hour infusion repeated after 12 hours (2 doses) on Day 2 in 21-day cycles.
Period: Overall Study
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Started | 80 | 52 | 55
Completed | 0 | 0 | 1
Not Completed | 80 | 52 | 54
Not completed — Lost to Follow-up | 3 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 3 | 0
Not completed — Death | 24 | 22 | 18
Not completed — Other | 45 | 27 | 35

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat population included all participants who were randomized into the study.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP | TOTAL
Number analyzed (Participants) | 80 | 52 | 55 | 187
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 56.4 (12.3) | 56.9 (11.4) | 55.9 (11.6) | 56.4 (11.8)
Age, Customized [Count of Participants; unit: Participants]
  < 65 YEARS | 60 | 35 | 43 | 138
  >= 65 YEARS | 20 | 17 | 12 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 19 | 24 | 78
  Male | 45 | 33 | 31 | 109

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate is defined as the proportion of participants with a best response of complete response (CR) or partial response (PR) according to the International Working Group criteria. CR is defined as disappearance of all evidence of disease. PR is defined as 50 percent (%) decrease in the sum of the product of the perpendicular diameters (SPD) of up to 6 largest dominant nodal masses and greater than or equal to (>=) 50% decrease in SPD of spleen/liver nodules.
Time Frame: From treatment administration (Day 1) to 90 days after the end of study treatment (up to approximately 36 months from the randomization of last participant)
Population: Intent-To-Treat population included all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 80 | 52 | 55
Percentage of participants | 47.5 [36.2 to 59.0] | 46.2 [32.2 to 60.5] | 43.6 [30.3 to 57.7]
Statistical Analysis 1: Comparison: Rituximab+ ICE/DHAP vs MEDI-551 4 mg/kg + ICE/DHAP; Test type: Superiority or Other; p = 0.5543, Cochran-Mantel-Haenszel

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from randomization until the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first according to the International Working Group criteria. PD is defined as appearance of any new lesions or >= 50% increase in SPD of more than one node or >= 50% increase in longest diameter of a previously identified node or >50% increase from nadir in the SPD of any previous lesions. PFS (months) = (Date of PD/death or censoring - Date of randomization + 1) / (365.25/12).
Time Frame: as for outcome 1
Population: Intent-To-Treat population included all participants who were randomized into the study.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 80 | 52 | 55
months | 6.1 [0.0 to 39.2] | 6.6 [0.0 to 31.3] | 7.7 [0 to 14.8]
Statistical Analysis 1: Comparison: Rituximab+ ICE/DHAP vs MEDI-551 4 mg/kg + ICE/DHAP; Test type: Superiority or Other; p = 0.8567, Log Rank

3. Secondary Outcome: Event-Free Survival (EFS)
Description: Event-Free Survival (EFS) is defined as the time from randomization until the first documentation of EFS events which include PD, initiation of alternative antitumor treatment or death due to any cause, whichever occurs first according to the International Working Group criteria. PD is defined as appearance of any new lesions or >= 50% increase in SPD of more than one node or >= 50% increase in longest diameter of a previously identified node or >50% increase from nadir in the SPD of any previous lesions. EFS (months) = (Date of EFS or censoring - Date of randomization + 1) / (365.25/12).
Time Frame: as for outcome 1
Population: Intent-To-Treat population included all participants who were randomized into the study.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 80 | 52 | 55
months | 4.7 [0.0 to 39.2] | 4.2 [0.0 to 31.3] | 5.9 [0.0 to 14.8]
Statistical Analysis 1: Comparison: Rituximab+ ICE/DHAP vs MEDI-551 4 mg/kg + ICE/DHAP; Test type: Superiority or Other; p = 0.7412, Log Rank

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death due to any cause according to the International Working Group criteria. OS (months) = (Date of death or censoring - Date of randomization + 1) / (365.25/12).
Time Frame: as for outcome 1
Population: Intent-To-Treat population included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 80 | 52 | 55
months | NA [15.6 to NA] — NA indicates data not estimable. | NA [14.2 to NA] — NA indicates data not estimable. | 23.0 [12.8 to NA] — NA indicates data not estimable.
Statistical Analysis 1: Comparison: Rituximab+ ICE/DHAP vs MEDI-551 4 mg/kg + ICE/DHAP; Test type: Superiority or Other; p = 0.9996, Log Rank

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression (TTP) is defined as the time from randomization until the first documentation of PD according to the International Working Group criteria. PD is defined as appearance of any new lesions or >= 50% increase in SPD of more than one node or >= 50% increase in longest diameter of a previously identified node or >50% increase from nadir in the SPD of any previous lesions. TTP (months) = (Date of PD or censoring - Date of randomization + 1) / (365.25/12).
Time Frame: as for outcome 1
Population: Intent-To-Treat population included all participants who were randomized into the study.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 80 | 52 | 55
months | 4.9 [0.0 to 11.1] | 4.2 [0.0 to 31.3] | 5.9 [0.0 to 14.0]
Statistical Analysis 1: Comparison: Rituximab+ ICE/DHAP vs MEDI-551 4 mg/kg + ICE/DHAP; Test type: Superiority or Other; p = 0.1686, Log Rank

6. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) is defined as the time from randomization until the first documentation of disease response according to the International Working Group criteria. Only participants who have achieved objective response (confirmed CR or confirmed PR) assessed by investigator were evaluated for TTR. CR is defined as disappearance of all evidence of disease. PR is defined as 50% decrease in the SPD of up to 6 largest dominant nodal masses and >= 50% decrease in SPD of spleen/liver nodules. TTR (months) = (Date of first disease response - Date of randomization + 1) / (365.25/12).
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized into the study. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 42 | 32 | 30
months | 1.7 [0.9 to 3.8] | 2.3 [1.5 to 3.4] | 2.3 [1.6 to 6.0]

7. Secondary Outcome: Duration of Response (DR)
Description: Duration of Response (DR) is defined as time from start of first documented objective response (confirmed CR or confirmed PR) to first documented PD according to the International Working Group criteria. CR is defined as disappearance of all evidence of disease. PR is defined as 50% decrease in the SPD of up to 6 largest dominant nodal masses and >= 50% decrease in SPD of spleen/liver nodules. PD: appearance of any new lesions or >= 50% increase in SPD of more than one node or >= 50% increase in longest diameter of a previously identified node or > 50% increase from nadir in the SPD of any previous lesions. Only participants who have achieved objective response assessed by investigator were evaluated. DR calculated as (months) = (Date of PD or censoring - Date of first disease response + 1)/ (365.25/12).
Time Frame: as for outcome 1
Population: Intent-To-Treat population included all participants who were randomized into the study. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 42 | 32 | 30
months | NA [4.9 to NA] — NA indicates data not estimable. | 7.1 [4.1 to NA] — NA indicates data not estimable. | 7.9 [4.6 to 12.2]

8. Secondary Outcome: Number of Participants With Best Overall Response Assessed by Blinded Independent Central Review (BICR)
Description: The best overall response was calculated, based upon the disease assessments recorded during the study visits, and summarized with the number of participants for the following categories: CR, PR, stable disease (SD), PD, and unknown. Responses were assessed according to the International Working Group criteria. CR: disappearance of all evidence of disease; PR: 50% decrease in the SPD of up to 6 largest dominant nodal masses and >= 50% decrease in SPD of spleen/liver nodules; PD: appearance of any new lesions or >= 50% increase in SPD of more than one node or >= 50% increase in longest diameter of a previously identified node or >50% increase from nadir in the SPD of any previous lesions; SD: failure to attain CR/PR or PD.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 80 | 52 | 55
Participants
  COMPLETE RESPONSE (CR) | 20 [16.0 to 35.9] | 6 [4.4 to 23.4] | 12 [11.8 to 35.0]
  PARTIAL RESPONSE (PR) | 18 | 18 | 12
  STABLE DISEASE (SD) | 17 | 12 | 14
  PROGRESSIVE DISEASE (PD) | 5 | 5 | 5
  UNKNOWN | 20 | 11 | 12

9. Secondary Outcome: Acceptable Dose of MEDI-551
Description: Acceptable dose for MEDI-551 was evaluated based on the benefit-risk analysis.
Time Frame: After the administration of the first dose of MEDI-551 (7 days before the Cycle 1) to last dose of MEDI-551 (Cycle 3 Day 1) (each cycle of 21 days)
Population: All participants who were randomized into the study and received MEDI-551.
Measure: Number; unit: milligram per kilogram (mg/kg)
Groups:
- MEDI-551: Participants were received MEDI-551 2 mg/kg or 4 mg/kg by IV infusion. Recommended MEDI-551 dose was selected based on the DMC reviews.
Arm/Group | MEDI-551
Number analyzed (Participants) | 107
milligram per kilogram (mg/kg) | 4

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended signs, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. Serious adverse event (SAE) is any AE that resulted in death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, life-threatening, a congenital anomaly/birth defect, or an important medical event. TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 90 days after the end of treatment (EOT).
Time Frame: as for outcome 1
Population: Safety population included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 79 | 52 | 54
Participants
  TEAEs | 78 | 51 | 52
  TESAEs | 33 | 25 | 27

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Hematology/Coagulation Laboratory Results
Description: An abnormal laboratory finding that was judged by the investigator to be clinically significant was reported as an AE. TEAEs were defined as events present at baseline that worsened in intensity after administration of MEDI-551, or events absent at baseline that emerged after administration of MEDI-551, for the period extending to 90 days after the end of study treatment (EOT).
Time Frame: as for outcome 1
Population: Safety population included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 79 | 52 | 54
Participants
  Anaemia | 47 | 32 | 33
  Febrile neutropenia | 16 | 9 | 12
  Granulocytopenia | 3 | 0 | 2
  Leukopenia | 9 | 6 | 10
  Lymphopenia | 4 | 2 | 3
  Neutropenia | 30 | 15 | 20
  Pancytopenia | 2 | 0 | 3
  Thromobocytopenia | 49 | 24 | 29
  Activated partial thromboplastin time prolonged | 0 | 2 | 0
  Blood immunoglobulin g decreased | 0 | 1 | 0
  Blood immunoglobulin m decreased | 0 | 1 | 0
  Haemoglobin decreased | 0 | 1 | 0
  Immunoglobulins decreased | 0 | 1 | 0
  Lymphocyte count decreased | 9 | 4 | 3
  Neutrophil count decreased | 7 | 6 | 8
  Platelet count decreased | 12 | 8 | 10
  Platelet count increased | 0 | 1 | 0
  White blood cell count decreased | 6 | 5 | 6

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Chemistry Laboratory Results (Include Urinalysis)
Description: An abnormal laboratory findings that was judged by the investigator to be clinically significant was reported as an AE. TEAEs were defined as events present at baseline that worsened in intensity after administration of MEDI-551, or events absent at baseline that emerged after administration of MEDI-551, for the period extending to 90 days after the end of study treatment.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 79 | 52 | 54
Participants
  Hyperbilirubinaemia | 1 | 0 | 0
  Hypernatraemia | 3 | 1 | 1
  Hyperphosphataemia | 0 | 0 | 2
  Hypertriglyerideaemia | 1 | 0 | 0
  Hyperuricaemia | 5 | 4 | 1
  Hypoalbuminaemia | 3 | 4 | 3
  Hypocalcaemia | 11 | 6 | 7
  Hypoglycaemia | 1 | 1 | 1
  Hypokalaemia | 24 | 13 | 14
  Hypomagnesaemia | 17 | 6 | 11
  Hyponatraemia | 8 | 2 | 2
  Hypophosphataemia | 4 | 3 | 3
  Hypoproteinaemia | 0 | 0 | 1
  Alanine aminotransferase increased | 7 | 2 | 4
  Aspartate aminotransferase increased | 5 | 2 | 6
  Blood alkaline phosphatase increased | 2 | 0 | 1
  Blood bicarbonate decreased | 1 | 0 | 0
  Blood bilirubin increased | 1 | 1 | 1
  Blood chloride increased | 0 | 1 | 0
  Blood creatinine increased | 10 | 5 | 7
  Blood lactate dehydrogenase increased | 2 | 1 | 1
  Blood magnesium decreased | 2 | 0 | 0
  Blood potassium decreased | 2 | 0 | 0
  Blood uric acid decreased | 0 | 1 | 0
  Blood uric acid increased | 1 | 1 | 0
  Gamma-glutamyltransferase increased | 9 | 3 | 3
  Hepatic enzyme increased | 1 | 0 | 1
  Protein total decreased | 0 | 1 | 1
  Transaminases increased | 1 | 2 | 0
  Dysuria | 2 | 1 | 3
  Hematuria | 2 | 3 | 0
  Glucose urine present | 0 | 1 | 1
  Proteinuria | 0 | 1 | 1
  Urine sodium increased | 0 | 0 | 1
  Calcium deficiency | 0 | 0 | 1
  Electrolyte imbalance | 2 | 0 | 0
  Hypercalcaemia | 2 | 1 | 0
  Hyperglycaemia | 12 | 9 | 2
  Hyperkalaemia | 2 | 2 | 1
  Hypermagnesaemia | 3 | 2 | 0

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Vital Signs and ECG Abnormalities
Description: Vital signs included parameters such as heart rate, blood pressure, temperature, and respiratory rate. An abnormal vital signs and ECG findings that was judged by the investigator to be clinically significant was reported an AE. TEAEs were defined as events present at baseline that worsened in intensity after administration of MEDI-551, or events absent at baseline that emerged after administration of MEDI-551, for the period extending to 90 days after the end of study treatment.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 79 | 52 | 54
Participants
  Arrhythmia | 0 | 0 | 2
  Atrial fibrillation | 1 | 1 | 2
  Bradycardia | 3 | 1 | 2
  Extrasystoles | 0 | 1 | 0
  Palpitations | 2 | 1 | 0
  Sinus arrhythmia | 0 | 0 | 1
  Sinus bradycardia | 1 | 2 | 1
  Systolic dysfunction | 0 | 0 | 1
  Tachycardia | 3 | 1 | 2
  Pyrexia | 17 | 14 | 11
  Blood pressure increased | 0 | 0 | 1
  Carbon dioxide decreased | 1 | 0 | 0
  Electrocardiogram abnormal | 0 | 0 | 1
  Electrocardiogram QT prolonged | 0 | 2 | 2
  Heart rate irregular | 1 | 0 | 0
  Weight decreased | 0 | 1 | 1
  Weight increased | 1 | 0 | 1
  Dyspnoea | 11 | 7 | 8
  Dyspnoea exertional | 0 | 3 | 1
  Hypertension | 5 | 2 | 3
  Hypotension | 10 | 4 | 8

14. Secondary Outcome: Number of Participants Who Developed Detectable MEDI-551 Anti-drug Antibodies (ADA)
Description: A participant was considered ADA-positive across the study if they had a positive reading (titer of 50 or higher) at any time point during the study.
Time Frame: 7 days before the start of Cycle 1, Day 1 of each subsequent Cycle, EOT, and post EOT on Days 30, 60, 90 and 270 (up to 36 months from the randomization of last participant)
Population: Safety population included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 52 | 54
Participants | 1 | 0

15. Secondary Outcome: Mean Serum Concentration of MEDI-551
Description: The mean serum concentration of MEDI-551 were observed.
Time Frame: Cycle 1 Day -7 Post dose, pre-dose and postdose on Day 1, post-dose on Days 4, 8, 15 of Cycle 1, pre-dose and postdose on Day 1 of Cycle 2 and Cycle 3
Population: Participants who received MEDI-551 were analyzed for this end point.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 52 | 54
mcg/mL
  Cycle 1 Day-7 Post Dose: number analyzed (Participants) | 46 | 50
  Cycle 1 Day-7 Post Dose | 47.0 (23.7) | 83.8 (21.9)
  Cycle 1 Day 1 Pre Dose: number analyzed (Participants) | 46 | 52
  Cycle 1 Day 1 Pre Dose | 16.7 (5.81) | 33.1 (16.3)
  Cycle 1 Day 1 Post Dose: number analyzed (Participants) | 46 | 51
  Cycle 1 Day 1 Post Dose | 64.8 (26.4) | 116 (41.3)
  Cycle 1 Day 4: number analyzed (Participants) | 43 | 45
  Cycle 1 Day 4 | 38.8 (14.6) | 71.9 (23.0)
  Cycle 1 Day 8: number analyzed (Participants) | 44 | 48
  Cycle 1 Day 8 | 30.6 (9.69) | 69.3 (25.1)
  Cycle 1 Day 15: number analyzed (Participants) | 40 | 43
  Cycle 1 Day 15 | 19.4 (6.19) | 44.7 (25.0)
  Cycle 2 Day 1 Pre Dose: number analyzed (Participants) | 40 | 44
  Cycle 2 Day 1 Pre Dose | 15.0 (5.45) | 30.9 (14.3)
  Cycle 2 Day 1 Post Dose: number analyzed (Participants) | 40 | 43
  Cycle 2 Day 1 Post Dose | 52.3 (18.7) | 112 (32.6)
  Cycle 3 Day 1 Pre Dose: number analyzed (Participants) | 26 | 26
  Cycle 3 Day 1 Pre Dose | 14.0 (6.50) | 36.4 (18.7)
  Cycle 3 Day 1 Post Dose: number analyzed (Participants) | 25 | 25
  Cycle 3 Day 1 Post Dose | 52.4 (16.9) | 116 (30.9)

16. Secondary Outcome: Half-life (T1/2) of MEDI-551
Description: Terminal elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: Cycle 1 and EOT (Day 21 of Cycle 3 [each cycle of 21 days] or earlier cycles if treatment stopped before Cycle 3)
Population: Participants who received MEDI-551 were analyzed for this end point.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Number analyzed (Participants) | 52 | 54
Day
  Cycle 1: number analyzed (Participants) | 36 | 43
  Cycle 1 | 14.4 (5.09) | 16.5 (10.5)
  End of Treatment: number analyzed (Participants) | 9 | 17
  End of Treatment | 18.9 (4.34) | 20.2 (5.73)

ADVERSE EVENTS:
Time Frame: From treatment administration (Day 1) to 90 days after the end of study treatment (up to approximately 36 months from the randomization of last participant)
Description: AE were reported for safety population, which included all participants who received any study treatment..
Arm/Group | Rituximab+ ICE/DHAP | MEDI-551 2 mg/kg + ICE/DHAP | MEDI-551 4 mg/kg + ICE/DHAP
Serious Adverse Events (participants affected / at risk) | 33/79 | 25/52 | 27/54
Other Adverse Events (participants affected / at risk) | 78/79 | 49/52 | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab+ ICE/DHAP (N=79) | MEDI-551 2 mg/kg + ICE/DHAP (N=52) | MEDI-551 4 mg/kg + ICE/DHAP (N=54)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11) | 8 (10) | 9 (10)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 1 (2) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 4 (5)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Coma hepatic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab+ ICE/DHAP (N=79) | MEDI-551 2 mg/kg + ICE/DHAP (N=52) | MEDI-551 4 mg/kg + ICE/DHAP (N=54)
Anaemia (Blood and lymphatic system disorders) | 47 (113) | 32 (87) | 33 (111)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 3 (4)
Granulocytopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 8 (10) | 6 (8) | 10 (31)
Lymphopenia (Blood and lymphatic system disorders) | 4 (22) | 2 (18) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 27 (50) | 15 (30) | 18 (45)
Thrombocytopenia (Blood and lymphatic system disorders) | 47 (172) | 24 (71) | 28 (114)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 0 (0) | 3 (3)
Dry eye (Eye disorders) | 4 (4) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 6 (9) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 23 (38) | 17 (23) | 18 (27)
Diarrhoea (Gastrointestinal disorders) | 19 (26) | 15 (17) | 13 (16)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (8) | 0 (0) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 43 (75) | 23 (45) | 25 (42)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 26 (37) | 14 (28) | 14 (21)
Asthenia (General disorders) | 9 (12) | 12 (21) | 11 (15)
Chills (General disorders) | 6 (9) | 1 (1) | 2 (2)
Fatigue (General disorders) | 22 (32) | 20 (33) | 15 (20)
Mucosal inflammation (General disorders) | 7 (7) | 3 (3) | 3 (5)
Oedema (General disorders) | 5 (6) | 1 (2) | 2 (2)
Oedema peripheral (General disorders) | 10 (12) | 6 (9) | 5 (7)
Pyrexia (General disorders) | 17 (24) | 12 (16) | 9 (10)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Oral herpes (Infections and infestations) | 4 (5) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (10) | 3 (3) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 11 (32) | 7 (9) | 6 (6)
Alanine aminotransferase increased (Investigations) | 7 (13) | 2 (2) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 5 (11) | 2 (2) | 6 (13)
Blood creatinine increased (Investigations) | 10 (17) | 5 (8) | 7 (17)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 2 (2) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 9 (15) | 3 (8) | 3 (4)
Lymphocyte count decreased (Investigations) | 9 (27) | 4 (13) | 3 (7)
Neutrophil count decreased (Investigations) | 7 (8) | 5 (8) | 8 (16)
Platelet count decreased (Investigations) | 12 (31) | 8 (38) | 10 (23)
White blood cell count decreased (Investigations) | 6 (13) | 4 (9) | 6 (22)
Decreased appetite (Metabolism and nutrition disorders) | 12 (14) | 7 (7) | 8 (11)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (23) | 8 (22) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (5) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (31) | 6 (9) | 7 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 24 (50) | 13 (23) | 14 (28)
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 (37) | 6 (10) | 11 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (11) | 2 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (10) | 3 (4) | 3 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (15) | 2 (2) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (9) | 7 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (8) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (5) | 1 (1)
Dizziness (Nervous system disorders) | 11 (12) | 8 (10) | 7 (9)
Dysgeusia (Nervous system disorders) | 3 (3) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 14 (19) | 7 (7) | 8 (10)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 2 (2) | 2 (3)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 7 (8) | 5 (5) | 2 (2)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 8 (9) | 4 (4) | 8 (8)
Acute kidney injury (Renal and urinary disorders) | 1 (4) | 3 (5) | 4 (5)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (3) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (3) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (4) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 9 (12) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 7 (11) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (5) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (7) | 5 (7) | 8 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 4 (4)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 6 (8)
Hypertension (Vascular disorders) | 5 (9) | 2 (2) | 3 (10)
Hypotension (Vascular disorders) | 10 (12) | 3 (4) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.